CLINICAL TRIAL: NCT01437761
Title: Hemodialysis With the 2008 Sorbent System: A Pilot Evaluation of Different Treatment Prescriptions
Brief Title: Sorbent Treatment Prescriptions Pilot Study
Acronym: Sorb2
Status: Terminated | Type: Observational
Why Stopped: Change of Institutional Affliation & Funding Changes
Sponsor: Renal Research Institute (Other)
Collaborators: Renal Solutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 150-11
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- 2008 Sorbent system: Hemodialysis with the 2008 Sorbent system
  Interventions: Device: 2008 Sorbent System

INTERVENTIONS:
Device: 2008 Sorbent System — 2008 Sorbent System with dialysate flow rates (Qd) of 400 and 500 ml/min while maintaining a constant blood flow rate (Qb) and constant dialyzer (KoA).

SUMMARY:
This study will compare how well blood of renal failure patients is cleaned with the new 2008 Sorbent System using two different dialysate speeds.

DETAILED DESCRIPTION:
The "2008 Sorbent System" is a new type of hemodialysis machine that requires only about 2 gallons of dialysate for a treatment because it can turn used dialysate into fresh dialysate again by filtering it through a special cleaning cartridge (called a "sorbent"). This new machine is approved by the U.S. Food and Drug Administration to clean the blood of patients whose kidneys have failed.

This study will compare the degree of blood cleansing achieved with the new 2008 Sorbent System using two different speeds at which the dialysate runs through the dialysis machine. This will tell us if the faster speed really does provide better cleaning (and how much) with this new machine.

How well the blood of a patient is cleaned by this procedure is determined by several factors. For example, longer treatment times generally provide better blood cleansing. Higher speeds at which the cleaning fluid runs through the artificial kidney do, too.

Since the 2008 Sorbent System is a new machine (and in some ways different from standard hemodialysis machines), other aspects may be different, too, between the 2008 Sorbent System and regular hemodialysis machines. Specifically, this study looks at how well this new machine corrects the patients' acid-base status (a common requirement in these patients), what effect the treatment has on inflammation in the patients' blood, how the levels of important substances in the blood are influenced (acetate, sulfate, nitrate, carbon dioxide), and if cleaning fluid in the 2008 Sorbent System contains any substances that are not found in the cleaning fluid used by regular hemodialysis machines.

ELIGIBILITY:
Inclusion Criteria:

* age </=18 years
* end-stage renal disease (ESRD) patient on chronic high-flux hemodialysis for </= 6 months at time of enrollment
* well-functioning fistula, graft or catheter as hemodialysis access, achieving blood flow rates of >/= 300 mL/min
* ability to understand the English language

Exclusion Criteria:

* Pre-dialysis serum blood urea nitrogen (BUN) concentration below 30 mg/dL in the last three months
* Severe Coronary Heart Disease or Heart Failure (New York Heart Association class IV)
* Active Infections
* Hepatitis B
* Any other active infection that has required antibiotic treatment in the preceding eight weeks
* Pre-study lab values of any of the following (in the most recent routine lab work)
* Sodium - Na+ > 150 mmol/L, Na+ < 132 mmol/L
* Potassium - K+ > 6.5 mmol/L, K+ < 3.5 mmol/L
* Total Calcium - Ca > 12 mg/dL (3 mmol/L), total Ca < 7.2 mg/dL (1.8 mmol/L)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment Adequacy | 4 weeks
  spKt/V, eKt/V, and Std Weekly Kt/V (Kt/V = dialysis adequacy)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Yorkville Dialysis Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No